CLINICAL TRIAL: NCT03258281
Title: Effects of Evolocumab on Platelet Reactivity in Patients With Diabetes Mellitus After Elective Percutaneous Coronary Intervention
Brief Title: Effects of Evolocumab on Platelet Reactivity in Patients With Diabetes Mellitus
Acronym: ISS-DMII
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Inova Health Care Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 17-2639
Record Dates: First submitted 2017-06-29; First posted 2017-08-23 (Actual); Results first posted 2023-01-19 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2022-12

CONDITIONS: Diabetes Mellitus, Type 2; Dyslipidemia Associated With Type II Diabetes Mellitus; Percutaneous Coronary Intervention
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — evolocumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- evolocumab 420mg (Active Comparator): 75 subjects on optimal statin therapy undergoing elective PCI will receive evolocumab 420mg.
  Interventions: Drug: Evolocumab
- placebo (Placebo Comparator): 75 subjects on optimal statin therapy undergoing elective PCI will receive placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Evolocumab — Patients will receive evolocumab 420 mg administered subcutaneously
  Other Names: Repatha
  Arms: evolocumab 420mg
Drug: Placebo — Patients will receive placebo administered subcutaneously
  Arms: placebo

SUMMARY:
Prospective, single center, double-blind, randomized pharmacodynamic experimental study. The study will enroll 150 subjects with ASCVD on optimal statin therapy as per physician and Diabetes Mellitus (DM) undergoing elective Percutaneous Coronary Intervention (PCI). Eligible patients will be randomized for 30 day treatment to either 1) evolocumab 420 mg ; or 2) placebo.

DETAILED DESCRIPTION:
This is a double-blind randomized clinical trial of evolocumab versus placebo in patients with ASCVD and DM on clopidogrel and aspirin undergoing PCI. The study is aimed to assess

1. the effect of evolocumab therapy on platelet activation and reactivity;
2. the effect of evolocumab on biomarkers of platelet activation and inflammation.

Eligible patients will be randomized prior to start the PCI equally to either:

1. 420 mg evolocumab ; or
2. placebo. The randomized treatment will be administered in subcutaneous injections.

The laboratory assessments will be performed before (baseline), and 16-24 hours and 30-days after randomization.

Subject participation will be 30 days from the randomization.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes Mellitus
* Dyslipidemia
* Undergoing elective PCI

Exclusion Criteria:

* Patients with recent Acute Coronary Syndrome (≤1 month)
* Patients on dual antiplatelet treatment (DAPT) with ticagrelor or prasugrel
* Patients undergoing urgent/emergent PCI for stent thrombosis
* Severe acute or chronic medical or psychiatric condition
* Pregnancy
* Participation in another experimental clinical trial, without formal approval
* Unwillingness or inability to comply with the requirements of this protocol

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-10-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Inova Fairfax Hospital, Falls Church, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 31 participants were screened, 4 met eligibility and were randomized to the study treatment.
Groups:
- Evolocumab 420mg: Participants on optimal statin therapy undergoing elective percutaneous coronary intervention (PCI) will receive evolocumab 420mg.
  Evolocumab: Participants will receive evolocumab 420 mg administered subcutaneously
- Placebo: Participants on optimal statin therapy undergoing elective percutaneous coronary intervention (PCI) will receive placebo
  Placebo: Participants will receive placebo administered subcutaneously
Period: Overall Study
Arm/Group | Evolocumab 420mg | Placebo
Started | 3 | 1
Completed | 3 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Evolocumab 420mg: Participants on optimal statin therapy undergoing elective PCI will receive evolocumab 420mg.
  Evolocumab: Participants will receive evolocumab 420 mg administered subcutaneously
- Placebo: Participants on optimal statin therapy undergoing elective PCI will receive placebo
  Placebo: Participants will receive placebo administered subcutaneously
- Total: Total of all reporting groups
Arm/Group | Evolocumab 420mg | Placebo | Total
Number analyzed (Participants) | 3 | 1 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (8) | 67 (0) | 69 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 1 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Adenosine Diphosphate (ADP) Stimulated P-selectin Expression
Description: Change from baseline in ADP-stimulated P-selectin expression (% Positive Cells) as measured by flow cytometry between treatment groups (420 mg evolocumab treatment and placebo).
Time Frame: Baseline and after 30 days of treatment
Population: Instrument malfunction with flow cytometer. Unable to collect data from subject (n=1) in placebo group.
Measure: Mean (Standard Deviation); unit: % Positive Cells
Arm/Group | Evolocumab 420mg | Placebo
Number analyzed (Participants) | 3 | 0
% Positive Cells
  Baseline | 45.2 (17.1) |
  30 Days | 47.8 (18.8) |

2. Secondary Outcome: Change in ADP-unstimulated P-selectin Expression
Description: Change in ADP-unstimulated P-selectin expression (% Positive Cells) between treatment groups (420 mg evolocumab treatment and placebo)
Time Frame: Baseline and after 30 days of treatment
Population: Instrument malfunction with flow cytometer. Unable to collect data from subject (n=1) in placebo group.
Measure: Mean (Standard Deviation); unit: % Positive Cells
Arm/Group | Evolocumab 420mg | Placebo
Number analyzed (Participants) | 3 | 0
% Positive Cells
  Baseline | 5.4 (2.7) |
  30 Days | 8.8 (2.9) |

3. Secondary Outcome: Change in ADP-stimulated Lectin-like oxLDL [Oxidized Low-density Lipoprotein] Receptor-1 Mean Fluorescence Intensity (MFI)
Description: Change in ADP-stimulated LOX-1 (MFI) as measured by flow cytometry between treatment groups (420 mg evolocumab treatment and placebo)
Time Frame: Baseline and after 30 days of treatment
Population: Instrument malfunction with flow cytometer. Unable to collect data from subject (n=1) in placebo group.
Measure: Mean (Standard Deviation); unit: MFI
Arm/Group | Evolocumab 420mg | Placebo
Number analyzed (Participants) | 3 | 0
MFI
  Baseline | 1186 (1017) |
  30 Days | 721 (82) |

4. Secondary Outcome: Change in ADP-stimulated Cluster of Differentiation (CD)-147 MFI
Description: Change in ADP-stimulated CD-147 mean fluorescence intensity (MFI) as measured by flow cytometry between treatment groups (420 mg evolocumab treatment and placebo)
Time Frame: Baseline and after 30 days of treatment
Population: Instrument malfunction with flow cytometer. Unable to collect data from subject (n=1) in placebo group.
Measure: Mean (Standard Deviation); unit: MFI
Arm/Group | Evolocumab 420mg | Placebo
Number analyzed (Participants) | 3 | 0
MFI
  Baseline | 1459 (1220) |
  30 Days | 678 (148) |

ADVERSE EVENTS:
Time Frame: 30 Days
Description: Any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product which does not necessarily have to have a causal relationship with this treatment. An adverse event can be any unfavorable and unintended sign symptom, or disease temporally associated with the use of a drug. This includes any newly occurring event that has increased in severity or frequency since the administration of the study treatment.
Arm/Group | Evolocumab 420mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/1
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/1
Other Adverse Events (participants affected / at risk) | 1/3 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Evolocumab 420mg (N=3) | Placebo (N=1)
Chest pain (Cardiac disorders) | 1 (1) | 0 (0) — Chest pain requiring hospitalization
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Evolocumab 420mg (N=3) | Placebo (N=1)
rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Study was terminated early as a result of 1) low enrollment and , 2) thrombosis research center moving to another health system (LifeBridge Health) . Only 4 patients were enrolled, as a result we were not able to conduct an analysis on any of the endpoints.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-04-24): https://cdn.clinicaltrials.gov/large-docs/81/NCT03258281/Prot_SAP_000.pdf
  • Informed Consent Form (2019-06-19): https://cdn.clinicaltrials.gov/large-docs/81/NCT03258281/ICF_001.pdf